CLINICAL TRIAL: NCT00631852
Title: A Phase II Biomarker Trial of Gelatin Encapsulated Extract of American Ginseng Root (LEAG) in Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Southern Illinois University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PER-SCCI 07-001.1
Record Dates: First submitted 2008-02-26; First posted 2008-03-10 (Estimated); Results first posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer, Biomarkers, Ginseng Root
MeSH Terms: conditions — Breast Neoplasms | interventions — Asian ginseng

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- American Ginseng root (Experimental): four, 250mg tablets daily 5-14 days prior to surgery
  Interventions: Drug: American Ginseng root

INTERVENTIONS:
Drug: American Ginseng root — four, 250mg tablets daily 5-14 days prior to surgery
  Other Names: LEAG; Ginseng

SUMMARY:
This study was designed to explore the changes brought about by gelatin encapsulated extract of American Ginseng Root (LEAG) in breast cancer tumors and surrounding normal breast epithelial cells. Various tumor biomarkers, as well as inflammatory mediators, will be examined in tissue following LEAG treatment.

DETAILED DESCRIPTION:
Asian ginseng (Panax ginseng) and its close relative American ginseng (Panax quinquefolium) are perennial aromatic herbs that are widely used in Asian medicine. Ginseng root is used as a tonic thought to increase the body's resistance to stress and fatigue, to increase endurance under heavy physical activity, and to improve well-being in age-related debilitation. Most of the ginseng consumed, even in Asian populations, is American ginseng, and the majority of American ginseng is grown and processed in Wisconsin, with quality and standardization overseen by the Ginseng Board of Wisconsin. Furthermore, in Asian medicine, Asian ginseng (Panax ginseng) and American ginseng (Panax quinquefolium) are common components in herbals used for cancer prevention and treatment. Indeed, retrospective studies have shown that patients who consumed ginseng on a regular basis experienced cancers at a reduced rate, however, breast cancer was not considered. Ginseng has been used medicinally for over 2000 years and there are no substantiated serious adverse effects, and few, if any, non-serious adverse effects. The World Health Organization lists ginseng as a traditional medicine with very low toxicity. Clinical trials have also demonstrated an anti-hyperglycemic action of American ginseng. These studies utilized capsules containing dried, ground Ontario-grown P. qinquefolius L. root. The ground AG root preparation had an onset of action of 40 minutes. They found no significant increase in anti-hyperglycemic action after 40 minutes and no significant increase in anti-hyperglycemic action using 1 gram versus 3 gram dosing.

LEAG is a standardized preparation of lyophilized water-extract of American ginseng root in 250-mg gelatin capsules. The ginseng was purchased through the Ginseng Board of Wisconsin and the lyophilized extract has been certified for percentage of each and total ginsenoside content and screened for safe levels of minerals, metals, and pesticides by ConsumerLab.com, a leading testing service company of dietary supplements.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cytologically confirmed breast cancer with biopsy showing invasive or non-invasive (DCIS) at least 1.0 cm greatest diameter on imaging
* Surgical patients undergoing lumpectomy, subtotal or total mastectomy
* 18 years of age or greater
* female
* available tissue blocks from diagnostic biopsy
* negative pregnancy test, medical history of surgical sterilization, or 1 year post menopausal
* must be willing to forego surgery for minimum of 5 days
* ability and willingness to sign written consent
* if hypertensive, on stable dose of medication at least 30 days
* if diabetic, well controlled (HbA1C < 8.5 within past 60 days or documented FPG < 140 mg/dl for 3 consecutive days
* ECOG status < 2 or Karnofsky of 60% or greater

Exclusion Criteria:

* previous or current malignancy, excluding non-melanomic skin cancer
* evidence of distant metastatic disease
* history of chemotherapy, biologic or radiotherapy with 6 months of biopsy
* usage of herbal supplements or alternative medications not approved by the FDA within 1 week of starting study drug. LEAG or related ginseng products, and combination products containing ginseng, should be discontinued within 6 weeks of starting study drug
* history of allergic reactions attributed to compounds of similar chemical or biologic composition to LEAG
* history of chronic inflammatory process, including, but not limited to, rheumatoid arthritis and lupus. This includes patients on concurrent systemic steroids or anti-inflammatory medications
* active bleeding or a pathological condition that carries a high risk of bleeding
* any swallowing dysfunction
* uncontrolled intercurrent illness
* poorly controlled diabetes (control indicated with HbA1c < 8.5 within past 60 days or documented fasting blood glucose < 140 mg/dl for three consecutive days)
* known diabetics who have experienced episodes of symptomatic hypoglycemia in the last 6 months are also considered poorly controlled and will be excluded from study participation.
* uncontrolled hypertension (SBP > 140 mmHg or DBP > 90 mmHG)
* pregnant or breast feeding women Women must be willing to use birth control throughout study duration.
* current investigational medications or treatment with an investigational agent within 6 weeks prior to biopsy
* current coumadin therapy or who have been treated with coumadin within the 2 weeks prior to biopsy
* current monoamine oxidase inhibitors treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-02; Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Peralta, M.D., Principal Investigator — Sutter Health
Locations (1):
- Simmons Cancer Institute-SIU School of Medicine, Springfield, Illinois, United States

REFERENCES:
- [Background] Peralta EA, Murphy LL, Minnis J, Louis S, Dunnington GL. American Ginseng inhibits induced COX-2 and NFKB activation in breast cancer cells. J Surg Res. 2009 Dec;157(2):261-7. doi: 10.1016/j.jss.2009.05.011. Epub 2009 Jun 6. PMID 19815237
- [Background] Peralta EA, Brewer AT, Louis S, Dunnington GL. Vitamin E increases biomarkers of estrogen stimulation when taken with tamoxifen. J Surg Res. 2009 May 1;153(1):143-7. doi: 10.1016/j.jss.2008.03.030. Epub 2008 Apr 22. PMID 18468636
- [Background] Peralta EA, Viegas ML, Louis S, Engle DL, Dunnington GL. Effect of vitamin E on tamoxifen-treated breast cancer cells. Surgery. 2006 Oct;140(4):607-14; discussion 614-5. doi: 10.1016/j.surg.2006.07.007. Epub 2006 Sep 6. PMID 17011908

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | American Ginseng Root
Started | 16 (Seventeen subjects were consented and 16 were considered enrolled and treated under the protocol. One was a screen fail.)
Completed | 16 (2 patients were administratively withdrawn after treatment had been completed as they declined sharing of data after PI transfer.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Platelet assay limited to 5 subjects per protocol. Serum markers limited to 11 subjects due to transfer of specimens to PI at new Institution. Not all subjects provided permission for transfer.
Arm/Group | American Ginseng Root
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16
Platelet Function Assay (PFA-100) [Mean (Full Range); unit: seconds] — Population: The first 5 patients enrolled had platelet function assessed prior to surgery with an interim analysis of platelet function and bleeding complications prior to additional patient enrollment to determine if platelet function should be evaluated in all study patients. After 5 patients completed the study protocol, a safety meeting was convened and determined that pre-operative platelet function assessment was not needed in all study patients.
  seconds
    number analyzed (Participants) | 5
    (all) | 142.8 [104 to 160]
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.3 (7.7)
Glucose [Mean (Full Range); unit: mg/dL] | 82 [61 to 108]
Estrogen Receptor Positivity [Count of Participants; unit: Participants] — Population: Data analyzed at a later date due to funding issues and PI transfer to new Institution. PI obtained funding through new Institution and only 11 subjects' approved transfer of source documents to new Institution.
  Participants
    number analyzed (Participants) | 11
    (all) | 7
Progesterone Receptor Positivity [Count of Participants; unit: Participants] — Population: ata analyzed at a later date due to funding issues and PI transfer to new Institution. PI obtained funding through new Institution and only 11 subjects' approved transfer of source documents to new Institution.
  Participants
    number analyzed (Participants) | 11
    (all) | 5
HER 2 Positivity [Count of Participants; unit: Participants] — Population: ata analyzed at a later date due to funding issues and PI transfer to new Institution. PI obtained funding through new Institution and only 11 subjects' approved transfer of source documents to new Institution.
  Participants
    number analyzed (Participants) | 11
    (all) | 1
Triple Negative Tumors [Count of Participants; unit: Participants] — Population: ata analyzed at a later date due to funding issues and PI transfer to new Institution. PI obtained funding through new Institution and only 11 subjects' approved transfer of source documents to new Institution.
  Participants
    number analyzed (Participants) | 11
    (all) | 4

OUTCOME MEASURES:

1. Primary Outcome: Adiponectin
Description: Change from baseline to completion of treatment with LEAG.
Time Frame: mean of 11.8 days
Population: Serum markers were analyzed at a later date due to funding issues and PI transfer to new Institution. PI obtained funding through new Institution and only 11 subjects' specimens were able to be transferred to new Institution.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | American Ginseng Root
Number analyzed (Participants) | 11
pg/ml | 1308 (11,985)

2. Primary Outcome: C Reactive Protein (CRP)
Description: Mean change from baseline to completion of treatment with LEAG.
Time Frame: mean of 11.8 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | American Ginseng Root
Number analyzed (Participants) | 11
pg/ml | 761 (1,347)

3. Primary Outcome: Hepatocyte Growth Factor (HGF)
Description: Mean change from baseline to completion of treatment with LEAG.
Time Frame: mean of 11.8 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | American Ginseng Root
Number analyzed (Participants) | 11
pg/ml | 1.25 (79.1)

4. Primary Outcome: Insulin Like Growth Factor 1 (IGF-1)
Description: Mean change from baseline to completion of treatment with LEAG.
Time Frame: mean of 11.8 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | American Ginseng Root
Number analyzed (Participants) | 11
pg/ml | -144 (478)

5. Primary Outcome: Insulin Like Growth Factor 1 Receptor (IGF-1R)
Description: Mean change from baseline following 10-14 days of treatment with LEAG.
Time Frame: 10-14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | American Ginseng Root
Number analyzed (Participants) | 11
pg/ml | -364 (1502)

6. Primary Outcome: Interlueken-1- (IL-10)
Description: Mean change from baseline to completion of treatment with LEAG.
Time Frame: mean 11.8 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | American Ginseng Root
Number analyzed (Participants) | 11
pg/ml | 0.1 (0.2)

7. Primary Outcome: IL-12p40
Description: Mean change from baseline to completion of treatment with LEAG.
Time Frame: mean 11.8 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | American Ginseng Root
Number analyzed (Participants) | 11
pg/ml | -1 (14)

8. Primary Outcome: IL-1b
Description: Mean change from baseline to completion of treatment with LEAG.
Time Frame: mean 11.8 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | American Ginseng Root
Number analyzed (Participants) | 11
pg/ml | 5 (13)

9. Primary Outcome: IL-1ra
Description: Mean change from baseline to completion of treatment with LEAG.
Time Frame: mean 11.8 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | American Ginseng Root
Number analyzed (Participants) | 11
pg/ml | 46 (687)

10. Primary Outcome: IL-2
Description: Mean change from baseline to completion of treatment with LEAG.
Time Frame: mean of 11.8 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | American Ginseng Root
Number analyzed (Participants) | 11
pg/ml | 2.7 (9.5)

11. Primary Outcome: IL-23
Description: Mean change from baseline to completion of treatment with LEAG.
Time Frame: mean 11.8 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | American Ginseng Root
Number analyzed (Participants) | 11
pg/ml | 26 (87)

12. Primary Outcome: IL-4
Description: Mean change from baseline to completion of treatment with LEAG.
Time Frame: mean 11.8 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | American Ginseng Root
Number analyzed (Participants) | 11
pg/ml | 29 (92)

13. Primary Outcome: IL-6
Description: Mean change from baseline to completion of treatment with LEAG.
Time Frame: mean 11.8 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | American Ginseng Root
Number analyzed (Participants) | 11
pg/ml | 4 (12)

14. Primary Outcome: IL-8
Description: Mean change from baseline to completion of treatment with LEAG.
Time Frame: mean 11.8 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | American Ginseng Root
Number analyzed (Participants) | 11
pg/ml | 1 (3)

15. Primary Outcome: Insulin
Description: Mean change from baseline to completion of treatment with LEAG.
Time Frame: mean 11.8 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | American Ginseng Root
Number analyzed (Participants) | 11
pg/ml | 299 (982)

16. Primary Outcome: Leptin
Description: Mean change from baseline to completion of treatment with LEAG.
Time Frame: mean 11.8 days
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: pg/ml
Arm/Group | American Ginseng Root
Number analyzed (Participants) | 11
pg/ml | -100 (438)

17. Primary Outcome: MCP-1
Description: Mean change from baseline to completion of treatment with LEAG.
Time Frame: mean 11.8 days
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: pg/ml
Arm/Group | American Ginseng Root
Number analyzed (Participants) | 11
pg/ml | 8 (20)

18. Primary Outcome: TGFb1
Description: Mean change from baseline to completion of treatment with LEAG.
Time Frame: mean 11.8 days
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: pg/ml
Arm/Group | American Ginseng Root
Number analyzed (Participants) | 11
pg/ml | 826 (3054)

19. Primary Outcome: TNFa
Description: Mean change from baseline to completion of treatment with LEAG.
Time Frame: mean 11.8 days
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: pg/ml
Arm/Group | American Ginseng Root
Number analyzed (Participants) | 11
pg/ml | -15 (51)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | American Ginseng Root
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 1/16
Other Adverse Events (participants affected / at risk) | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | American Ginseng Root (N=16)
hemorrhage/ bleeding (Blood and lymphatic system disorders) | 1 (1) — Pt had episode of increased bleeding in JP drain after mastectomy + reconstruction. Output >250mL over a 2 hours on post-op day 5. Pt returned to OR on post-op day 6 for evacuation of hematoma & discharged post op day 7. Resolved by post-op day 12.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | American Ginseng Root (N=16)
pain (General disorders) | 15 (15) — Pain at surgical incision site
numbness (Nervous system disorders) | 1 (1) — numbness in arm at surgical drain site.
syncope (General disorders) | 1 (1) — dizziness ann syncope
decreased sensation of digits (Nervous system disorders) | 1 (1) — lack of feeling in 2nd and 3rd digits bilaterally.
coolness in digits (Nervous system disorders) | 1 (1) — Coolness/ feeling cold in 2nd and 3rd digits bilaterally.
Floater in eye (Eye disorders) | 1 (1) — Visual sensation of a "floater" in right eye.
headache (General disorders) | 7 (7) — headache
back pain (General disorders) | 1 (1) — pain in back.
soar throat (Gastrointestinal disorders) | 1 (1) — pain in throat.
injection site reaction (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Injection site reaction resulting in airway obstruction from IV morphine sulfphate.
decreased oxygen saturation (Respiratory, thoracic and mediastinal disorders) | 2 (2) — O2 saturation dropped below 90%.
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) — shortness of breath as perceived by patient.
Edema (Blood and lymphatic system disorders) | 3 (3) — Edema of upper extremity following surgery.
edema (Surgical and medical procedures) | 2 (2) — Edema at surgical and reconstructive sites.
Fatigue (General disorders) | 3 (3) — Feeling of tiredness.
Hyperactivity (General disorders) | 2 (2) — Feeling of excessive energy and need to keep moving.
Fever (General disorders) | 1 (1)
hiccups (Gastrointestinal disorders) | 1 (1)
hot flash (General disorders) | 1 (1)
Insomnia (General disorders) | 2 (2)
nightmares (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-05): https://cdn.clinicaltrials.gov/large-docs/52/NCT00631852/Prot_SAP_000.pdf